CLINICAL TRIAL: NCT05319093
Title: Observational Study of the Effect of Ozanimod on Fatigue in Multiple Sclerosis Patients
Status: Terminated | Type: Observational
Why Stopped: Funding ended prematurely
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Charles Guttmann, MD, Director, Center for Neurological Imaging, Brigham and Women's Hospital
Other Study IDs: 2021P003284
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Fatigue; Multiple Sclerosis
Keywords: fatigue; multiple sclerosis; brain; ozanimod; diffusion MRI
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early Ozanimod treatment: In this group the effect of Ozanimod will be assessed in patients who initiated on Ozanimod treatment at study baseline (n=10).
  Treatment schedule and dosage of Ozanimod and the other disease-modifying treatments (DMTs) will be solely based on clinical indication and will be instituted by the patient's treating neurologist at Brigham and Women's Hospital or Massachusetts General Hospital.
  Interventions: Drug: Ozanimod
- Medium-term Ozanimod treatment: In this group, the effect of Ozanimod will be assessed in patients treated with Ozanimod for ≥6 months at study baseline (n=10).
  Treatment schedule and dosage of Ozanimod and the other disease-modifying treatments (DMTs) will be solely based on clinical indication and will be instituted by the patient's treating neurologist at Brigham and Women's Hospital or Massachusetts General Hospital.
  Interventions: Drug: Ozanimod
- Non-Ozanimod treatment: In this group, investigators will involve patients initiated on any disease-modifying drug (other than Ozanimod) at study initiation (n=10).
  Treatment schedule and dosage of the disease-modifying treatments (DMTs) will be solely based on clinical indication and will be instituted by the patient's treating neurologist at Brigham and Women's Hospital or Massachusetts General Hospital. The proposed study is purely observational and will not influence the selection, schedule or dosage of patient treatments.
- Untreated: In this group, MS patient will be involved who did not receive any disease-modifying drug for at least 3 months before study initiation (i.e., untreated patients, n=10)

INTERVENTIONS:
Drug: Ozanimod — Three-months, longitudinal observational period
  Other Names: ZEPOSIA
  Groups: Early Ozanimod treatment; Medium-term Ozanimod treatment

SUMMARY:
Multi-center observational study to assess the short-term response of multiple sclerosis (MS) patients initiated on Ozanimod with respect to fatigue. Patterns of brain changes on brain magnetic resonance imaging (MRI) that might modulate the effect of Ozanimod treatment on fatigue will also be assessed.

DETAILED DESCRIPTION:
Primary objectives:

1. To assess the effect of Ozanimod treatment on the impact of fatigue on physical, cognitive, and psychosocial functions, as measured by the modified fatigue impact scale (MFIS).
2. To assess the impact of fronto-striatal damage on the association between Ozanimod treatment and fatigue.

Secondary objectives:

1. To assess the effect of Ozanimod treatment on fatigue severity, mood symptoms (ie, depression and anxiety), sleep quality, physical activity, reward responsiveness and cognitive functions over the first 3-month after treatment initiation with Ozanimod.
2. To assess the time course of changes by daily administration of visual analogue scales of fatigue, depression, anxiety, and pain, and monthly administration of self-assessment questionnaires for fatigue, depression and anxiety using a mobile application.
3. In addition to the hypothesis-driven analyses specifically targeting the fronto-striatal system, the investigators will also perform analyses designed to discover other potential brain MRI predictors of Ozanimod treatment response (ie, change in primary and/or secondary endpoints during the 3-month Ozanimod treatment). The investigators will perform global and regional (e.g., cerebral cortical, deep grey matter, hippocampal) volumetric measurements as well as well-established voxel-based image statistics to seek other potential patterns of brain atrophy that identify responders to Ozanimod. Resting state functional MRI (rsfMRI) will also be performed to seek potential markers of fatigue related to functional brain connectivity changes.
4. To establish patient compliance in using the aforementioned mobile app, and the robustness of app-based phenotypic characterization of fatigue and related symptoms on real-world patients. These observations will lay the basis for future prospective studies on larger patient cohorts. For this purpose, recruitment will also be expanded to patients treated with disease modifying drugs other than Ozanimod.

Primary hypothesis:

Patients without significant damage to fronto-striatal circuitry (ie, fronto-striatal fractional anisotropy (FA)≥0.26 on diffusion tensor MRI (DT-MRI)) show significant decrease in fatigue score over the first 3-month after treatment initiation with Ozanimod.

Study assessments:

Treatment schedule and dosage of Ozanimod and the other disease-modifying treatments (DMTs) will be solely based on clinical indication and will be instituted by the patient's treating neurologist at Brigham and Women's Hospital or Massachusetts General Hospital. The proposed study is purely observational and will not influence the selection, schedule or dosage of patient treatments. Therefore, no safety assessment will be performed within the study.

All endpoints and confounders will be assessed using state-of-the art mobile/wearable technology, while the patient is on her/his/their normal routine at home and/or at work, including self-isolated quarantine. All patient-reported outcomes (PROs) will be assessed using a mobile application developed by the study team. The first version of the mobile application was already tested and used in a prospective brain MRI study of MS-related fatigue (MGB IRB Protocol number: 2017P001239). The mobile application will be modified and adapted to make it specifically suitable for the proposed study. The application will be installed on an Android smartphone that will be provided to each subject. The application will communicate using end-to-end encryption (https protocol) with a server inside the MGB firewall. Data will be transmitted between the mobile app and the server in deidentified and coded form.

Continuous actigraphy will be performed using wrist-worn actigraphic watches to assess quantitative physical activity (during daytime) and sleep measures (at night) during the entire 3-months period of the trial. These devices also measure other bio-signals as for instance skin conductivity and heart rhythm, as well as light exposure.

Presence/absence of obstructive sleep apnea and restless leg syndrome will be assessed once between day 0 and day 3 of the trial period using a home sleep test (HST) device.

Subjects will receive the study devices in person or via postal mail and will be instructed how to use the devices in person or via video conference call in compliance with COVID-19 regulations.

Each patient will undergo 3 Tesla brain Magnetic Resonance Imaging, including diffusion tensor, T1-weighted, T2-weighted, FLAIR and rsfMRI imaging at Brigham and Women's Hospital at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18
2. diagnosis of MS (according to the 2010 McDonald criteria)

Exclusion Criteria:

1. neurodegenerative disorders other than MS
2. terminal medical condition
3. currently treated for active malignancy
4. alcohol or substance abuse in the past year, except marijuana
5. non-English speakers (the mobile application is not available in other languages)
6. inability to undergo MRI scan

Patients undergoing COVID-19 vaccination will be allowed to participate in the study if at least 2 weeks have elapsed from their last dose of vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All MS patients seen at Brigham and Women's Hospital and Massachusetts General Hospital who fit our selection criteria (see below) will be eligible to participate in this study. Since MS is 2-3 times more common in women, investigators expect that more women than men will participate.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Three-months change in Modified Fatigue Impact Scale (MFIS) score | 3 months
  Difference in Modified Fatigue Impact Scale (MFIS) score between baseline (treatment initiation) and month 3. MFIS score will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period. Should the 84-day measurement not be available, the three-months change will be estimated by linear regression extrapolation using available measurements.

SECONDARY OUTCOMES:
Three-months change in Chalder Fatigue Scale (CFS) score | 3 months
  Difference in Chalder Fatigue Scale (CFS) score between baseline (treatment initiation) and month 3. CFS score will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period. Should the 84-day measurement not be available, the three-months change will be estimated by linear regression extrapolation using available measurements.
Three-months change in Fatigue Severity Scale (FSS) score | 3 months
  Difference in Fatigue Severity Scale (FSS) score between baseline (treatment initiation) and month 3. FSS score will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period. Should the 84-day measurement not be available, the three-months change will be estimated by linear regression extrapolation using available measurements.
Three-months change in NeuroQOL-fatigue questionnaire score | 3 months
  Difference in NeuroQOL-fatigue scale score between baseline (treatment initiation) and month 3. NeuroQOL-fatigue score will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period. Should the 84-day measurement not be available, the three-months change will be estimated by linear regression extrapolation using available measurements.
Visual Analog Scale (VAS) for fatigue score | 3 months
  Change in VAS fatigue score over the observation period. Current fatigue level will be assessed using VAS every four hours while the patient is awake during the trial period.
Three-months change in NeuroQOL-cognitive function questionnaire score | 3 months
  Difference in NeuroQOL-cognitive function scale score between baseline (treatment initiation) and month 3. Cognitive function will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period. Should the 84-day measurement not be available, the three-months change will be estimated by linear regression extrapolation using available measurements.

OTHER OUTCOMES:
NeuroQOL-depression scale | 3 months
  Level of depression will be assessed using the NeuroQOL-depression scale score. It will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period.
NeuroQOL-anxiety scale | 3 months
  Level of anxiety will be assessed using the NeuroQOL-anxiety scale score. It will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period.
Epworth Sleepiness scale | 3 months
  Sleep abnormalities will be assessed using the Epworth Sleepiness scale score. It will be assessed at baseline, as well as on days 28, 56 and 84 of the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Charles RG Guttmann, MD, Principal Investigator — Brigham and Women's Hospital, Radiology
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palotai M, Wallack M, Kujbus G, Dalnoki A, Guttmann C. Usability of a Mobile App for Real-Time Assessment of Fatigue and Related Symptoms in Patients With Multiple Sclerosis: Observational Study. JMIR Mhealth Uhealth. 2021 Apr 16;9(4):e19564. doi: 10.2196/19564. PMID 33861208
- [Background] Cella M, Chalder T. Measuring fatigue in clinical and community settings. J Psychosom Res. 2010 Jul;69(1):17-22. doi: 10.1016/j.jpsychores.2009.10.007. Epub 2009 Dec 11. PMID 20630259
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Cella D, Lai JS, Nowinski CJ, Victorson D, Peterman A, Miller D, Bethoux F, Heinemann A, Rubin S, Cavazos JE, Reder AT, Sufit R, Simuni T, Holmes GL, Siderowf A, Wojna V, Bode R, McKinney N, Podrabsky T, Wortman K, Choi S, Gershon R, Rothrock N, Moy C. Neuro-QOL: brief measures of health-related quality of life for clinical research in neurology. Neurology. 2012 Jun 5;78(23):1860-7. doi: 10.1212/WNL.0b013e318258f744. Epub 2012 May 9. PMID 22573626
- [Background] Palotai M, Guttmann CR. Brain anatomical correlates of fatigue in multiple sclerosis. Mult Scler. 2020 Jun;26(7):751-764. doi: 10.1177/1352458519876032. Epub 2019 Sep 19. PMID 31536461
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Palotai M, Weiner HL, Chitnis T, Duffy JF, and Guttmann CR, SLEEP APNEA AND PERIODIC LIMB MOVEMENTS ARE HIGHLY PREVALENT IN PATIENTS WITH MULTIPLE SCLEROSIS in 34th Annual Meeting of the Associated Professional Sleep Societies; Sleep, Volume 43, Issue Supplement_1, April 2020, Pages A429-A430, 1122. 2020.
- [Background] Billiard M, Broughton R. Modafinil: its discovery, the early European and North American experience in the treatment of narcolepsy and idiopathic hypersomnia, and its subsequent use in other medical conditions. Sleep Med. 2018 Sep;49:69-72. doi: 10.1016/j.sleep.2018.05.027. Epub 2018 Jun 6. PMID 30174215
- [Background] Miller P, Soundy A. The pharmacological and non-pharmacological interventions for the management of fatigue related multiple sclerosis. J Neurol Sci. 2017 Oct 15;381:41-54. doi: 10.1016/j.jns.2017.08.012. Epub 2017 Aug 12. PMID 28991714
- [Background] Yang TT, Wang L, Deng XY, Yu G. Pharmacological treatments for fatigue in patients with multiple sclerosis: A systematic review and meta-analysis. J Neurol Sci. 2017 Sep 15;380:256-261. doi: 10.1016/j.jns.2017.07.042. Epub 2017 Jul 28. PMID 28870581
- [Background] Induruwa I, Constantinescu CS, Gran B. Fatigue in multiple sclerosis - a brief review. J Neurol Sci. 2012 Dec 15;323(1-2):9-15. doi: 10.1016/j.jns.2012.08.007. Epub 2012 Aug 27. PMID 22935407
- [Background] Kos D, Kerckhofs E, Nagels G, D'hooghe MB, Ilsbroukx S. Origin of fatigue in multiple sclerosis: review of the literature. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):91-100. doi: 10.1177/1545968306298934. Epub 2007 Apr 4. PMID 17409388
- [Background] Palotai M, Cavallari M, Healy BC, Guttmann CR. A novel classification of fatigue in multiple sclerosis based on longitudinal assessments. Mult Scler. 2020 May;26(6):725-734. doi: 10.1177/1352458519898112. Epub 2020 Jan 23. PMID 31971067
- [Background] Palotai M, Cavallari M, Koubiyr I, Morales Pinzon A, Nazeri A, Healy BC, Glanz B, Weiner HL, Chitnis T, Guttmann CR. Microstructural fronto-striatal and temporo-insular alterations are associated with fatigue in patients with multiple sclerosis independent of white matter lesion load and depression. Mult Scler. 2020 Nov;26(13):1708-1718. doi: 10.1177/1352458519869185. Epub 2019 Aug 16. PMID 31418637
- [Background] Palotai M, Nazeri A, Cavallari M, Healy BC, Glanz B, Gold SM, Weiner HL, Chitnis T, Guttmann CRG. History of fatigue in multiple sclerosis is associated with grey matter atrophy. Sci Rep. 2019 Oct 14;9(1):14781. doi: 10.1038/s41598-019-51110-2. PMID 31611598
- [Background] Cavallari M, Palotai M, Glanz BI, Egorova S, Prieto JC, Healy BC, Chitnis T, Guttmann CR. Fatigue predicts disease worsening in relapsing-remitting multiple sclerosis patients. Mult Scler. 2016 Dec;22(14):1841-1849. doi: 10.1177/1352458516635874. Epub 2016 Feb 26. PMID 26920374
- [Background] Palotai M, Mike A, Cavallari M, Strammer E, Orsi G, Healy BC, Schregel K, Illes Z, Guttmann CR. Changes to the septo-fornical area might play a role in the pathogenesis of anxiety in multiple sclerosis. Mult Scler. 2018 Jul;24(8):1105-1114. doi: 10.1177/1352458517711273. Epub 2017 May 26. PMID 28548605
- See also: MotionWatch 8 — http://www.camntech.com/motionwatch-8/?gclid=CjwKCAjwu5CDBhB9EiwA0w6sLasykklM0I-K0nPtxe4WNO8wt4yV8m91jhcsbsbwHDVbSNfnBYuUVhoCpgQQAvD_BwE.
- See also: Nox T3s Home Sleep Device — http://noxmedical.com/noxt3s/?utm_term=nox%20t3%20sleep%20monitor&utm_campaign=%5BSearch%5D+Brand+-++Product+%5Be%5D&utm_source=adwords&utm_medium=ppc&hsa_acc=7911060515&hsa_cam=1382669894&hsa_grp=60659555971&hsa_ad=267498377165&hsa_src=g&hsa_tgt=kwd-422694661172&hsa_kw=nox%20t3%20sleep%20monitor&hsa_mt=e&hsa_net=adwords&hsa_ver=3&gclid=CjwKCAjwu5CDBhB9EiwA0w6sLQEnEeTrdfAzYAkRsa0tL5cQsoRGr3jaqz1GRp5jbfKeqDvZokx56RoCv8IQAvD_BwE